CLINICAL TRIAL: NCT04142138
Title: Translational Characterization of Blood Pressure Changes Following the Dietary Approach to Stop Hypertension (DASH) Diet- From Nutrition Through Electrolytes to Exosomes.
Brief Title: When the Kidney Reacts to Nutritional Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DBI-1000
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Prehypertension
Keywords: inpatient; nutrition
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Intervention Model Description: This study assesses how nutritional changes, namely DASH diet, change the composition of ion channels in the renal tubule, as exemplified by urine electrolyte ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nutrition implementation (Experimental): Volunteers with prehypertension, but otherwise healthy, will complete a screening visit, then be admitted to the In-Patient Unit for fourteen (14) days. Participants will be admitted for 5 days during the week and then go on pass for 2 weekend days each week with packed DASH diet meals. During hospitalization we will: 1) collect samples of blood and urine daily 2) monitor blood pressure, weight and pulse twice daily 3) collect 24-hour urine, twice during the period of two weeks 4) serve participants a menu based on DASH principles, namely low in sodium and high in potassium.
  Interventions: Other: DASH

INTERVENTIONS:
Other: DASH — DASH diet is based on low salt, high potassium components, and is comprised of mainly fruits and vegetables. During hospitalization we will collect laboratory data of blood and urine, and follow participants clinically by measuring blood pressure.

SUMMARY:
Hypertension is one of the leading causes of morbidity and mortality in the industrialized world, attributed mostly to modifiable lifestyle factors. Aspects that are controlled by patients include physical activity, smoking, alcohol consumption, and nutrition. The DASH (Dietary Approach to Stop Hypertension) diet is a proven effective intervention in lowering blood pressure in multiple populations. In this proof of concept study, volunteers with untreated stage 1 hypertension, defined as mild high blood pressure with numbers in the range of 130 - 139 over 80 - 89, will receive a DASH-based menu during 5 days of hospitalization, during a weekend at home where they will continue the menu, another 5 days as inpatients, followed by a weekend at home on the same menu, and the return to the inpatient unit for an additional day for final testing. Throughout the intervention period, participants will be followed clinically and undergo repeated laboratory testing. The aim of this project is to characterize changes in urine electrolytes and exosome protein abundance pattern during nutritional changes, shifting from a "westernized diet" to a DASH diet.

DETAILED DESCRIPTION:
Diet is a major disease modifier of hypertension. The Dietary Approaches to Stop Hypertension diet (DASH) is endorsed nationally and abroad to treat hypertension (HTN) in adults. In the original DASH study, the effect of the combination diet consisting of low salt, high potassium, and low-fat dairy products, was more pronounced in hypertensives and minorities. The magnitude of the effect on blood pressure (BP) of the combination diet was similar to that observed with single drug antihypertensive therapy.

Americans typically consume 3400 mg sodium daily, due to high intakes of processed foods, frequent eating outside the home, and consumption of packaged meals and salty snack foods. Foods consumed outside of the home provide 34% of the sodium intake of Americans.

It is not known exactly how the DASH diet effects its lowering of blood pressure. One of the proposed mechanism of the effect of the DASH diet relies on two components - sodium reduction and potassium supplementation.

In response to potassium supplementation such as in DASH diet, we would expect less sodium to be reabsorbed.

Over the years, adherence to DASH diet has been evaluated using questionnaires. Methods for monitoring sodium intake remain inadequate and flawed. Dietary recall is not reliable, and many patients truly do not realize, and consequently under report, the amount of sodium they consume. The most widely employed method of assessing dietary adherence, the 24-h urine collection to measure sodium excretion, is cumbersome and inconvenient. Evaluating urine sodium to creatinine ratio was validated as a surrogate measure to 24-hour urine collection .

Exosomes: most of the data regarding tissue activity of different channels in response to stimuli, comes from animal studies. Translation of the murine experimental findings to a human setting is difficult and has mostly been inferred using plasma and urinary electrolyte levels as a proxy for renal tubular transporter activity. Transporter proteins from all tubular segments are excreted into the urine in extracellular vesicles. These vesicles therefore provide a non-invasive liquid biopsy access to tubular epithelial cells that could potentially inform on physiological regulation of transporter activity in human kidneys . The proteins that are present in urine are a major area of investigation for proteomics researchers. In normal urine, typically half of the proteins are soluble proteins (49%), and the remaining 48% are sediment precipitated with low-speed centrifugation, and exosomes (3%). All exosomes contain a few common protein components. The cytosolic proteins present on exosomes include annexins, adhesion molecules, proteins that participate in vesicle formation and trafficking and metabolic enzymes. Analysis of urine exosomes can enhance the detectability of relatively low-abundant proteins that have potential pathophysiological significance, and so have become one of the newer trends in the field of urine-biomarker discovery .

Volunteers with hypertension stage 1, but otherwise healthy, will complete a screening visit, then be admitted to the In-Patient Unit for fourteen (14) days. Participants will be admitted for 5 days during the week and then go on pass for 2 weekend days each week with packed DASH diet meals. During hospitalization blood and urine samples will be collected daily, as well as clinical parameters such as blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. any gender, 18-60 years of age
2. self described as White or Black individuals
3. prehypertensives (=stage 1 hypertension) defined as sustolic blood pressure of 130-159 mmHG and/or diastolic blood pressure between 80-100.
4. adequate dentition to consume fruits and vegetables as described for DASH -

Exclusion Criteria:

1. Preexisting kidney disease structural or parenchymal including APCKD (adult polycystic kidney disease), single kidney (as assessed by ultrasound including size differences >3 cm in diameter between kidneys), or evidence of RAS (renal artery stenosis)
2. Pregnant
3. HIV
4. taking medications for diabetes, hyperlipidemia, cardiac disease, Medications for birth control, psychiatirc conditions, and sleep are Ok. Vitamins and herbs are Ok if continued throughout the study. Thyroid meds are acceptable if the TSH is within normal limits.
5. Diabetes as defined by hemoglobin A1c > 6.5% and/or fasting glucose > 125 mg/dl
6. Hyperlipidemia as defined by triglycerides >200 and/or LDL > 150
7. Hematuria on screening
8. RAAS (Renin-Angiotensin-Aldosterone) axis deviation - Aldosterone and Renin should be within normal ranges upon screening.
9. BUN > 40mg/dL corrected to body surface area
10. Creatinine > 1.3 mg/dL corrected to body surface area
11. BMI > 29.9 or < 19
12. Current smoker
13. Currently, a vegetarian (who does not consume fish and dairy) or a vegan
14. Based on medical history, any evidence of an autoimmune disease
15. Use of any of the following - ACEi, ARB, spironolactone, diuretics of any class, beta blockers, alpha blockers, nsaids, within the past two weeks
16. Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
urine exosome protein abundance pattern | Day 1 and Day 12
  Mass spectrometry generates a list of proteins for each sample. We will compare fold of change before (Day 1) and after intervention (Day 12) - a true change is defined as 1.5 fold.
urine electrolyte ratio in a spot urine as a surrogate to 24-h urine collection to assess nutritional consumption. | day 1,2,3,4,5,6,8,9,10,11,12,14
  spot urine will be analyzed for sodium and potassium parallel to 24-h urine collection. We will assess the concordance between the 24-h collection and the spot urine ratio of electrolytes. The result will be presented as a ratio of SPOT ratio (sodium/potassium) to 24-h collection ratio (sodium/potassium), for each participant. We will assess how close the ratio of ratios is to one.
24-h urine collection as a measure of adherence to the DASH diet | day 1, 12
  Urine will be collected throughout 24 hours to analyze electrolyte content, during intervention - twice, at the beginning (day 1) and end of intervention (day 12). We will be measuring daily sodium excretion, the threshold for compliance will be equal to or less than 100MEQ/d. For potassium daily excretion the threshold will be greater than or equal to 90meq/d . The change will be reported as number of participants that have met the defined threshold for compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Bielopolski, MD PhD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No